CLINICAL TRIAL: NCT04432376
Title: Randomized, Double-blind, Phase III Study of the Efficacy and Safety of Miconazole Oil Versus Vehicle Oil in the Treatment of Otomycosis, Followed by an Open-label Safety Evaluation
Brief Title: Efficacy and Safety Study of Miconazole Oil Versus Vehicle on Fungal Infection of the Ear Canal (Otomycosis)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hill Dermaceuticals, Inc. (Industry)
Collaborators: Abond CRO Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MZ-0120-ESP3-052
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Results first posted 2022-11-04 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Otomycosis
MeSH Terms: conditions — Otomycosis | interventions — Miconazole; Oils

STUDY DESIGN:
Intervention Model Description: Two phases; initial is randomized double-blind active vs placebo on a pre-determined number of subjects with otomycosis, to finish before starting second phase. Second phase is open-label use on diseased or healthy subjects to evaluate safety. Subjects from initial phase may crossover to second phase open-label if they meet the requirements, and new diseased or healthy subjects meeting requirements may enroll in this open-label phase.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Clinical Investigators, study staff and subjects randomized to the initial phase of the study are blinded to active drug and placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Active treatment arm (Active Comparator): Treatment with miconazole 2% oil, 5 drops into each ear twice daily for 14 consecutive days
  Interventions: Drug: miconazole 2% oil
- Placebo treatment arm (Placebo Comparator): Treatment with the vehicle oil, placebo, 5 drops into each ear twice daily for 14 consecutive days
  Interventions: Drug: vehicle oil
- Open-label treatment arm (Other): Application of miconazole 2% oil, 5 drops into each ear twice daily for 14 consecutive days
  Interventions: Drug: miconazole 2% oil

INTERVENTIONS:
Drug: miconazole 2% oil — Drug treatment of otomycosis for 14 days
  Other Names: active treatment
  Arms: Active treatment arm; Open-label treatment arm
Drug: vehicle oil — Placebo treatment of otomycosis for 14 days
  Other Names: placebo treatment
  Arms: Placebo treatment arm

SUMMARY:
This study involves two portions, a randomized, double-blind portion and an open-label portion, to evaluate the efficacy and safety of Miconazole oil 2% versus its Vehicle in the treatment of fungal infection of the outer ear canal (Otomycosis). The subjects randomized in the first portion of the study will have active fungal infection of the ear(s) and will be treated with either Miconazole Oil or the Vehicle for 14 days twice daily, 5 drops into the affected ear(s) per dose. The subjects enrolled in the open-label portion of the study may or may not have active fungal infection of the ear(s), and will be given the Miconazole Oil active drug following the same application of 5 drops into the ear(s) twice daily for 14 days.

The intention of the study is to evaluate the efficacy of Miconazole Oil on fungal infection of the ears when applied using 5 drops into the ear(s) twice daily for 14 days continuously. This study also intends to show safety of Miconazole Oil 5 drops into each ear twice a day for 14 consecutive days.

DETAILED DESCRIPTION:
This study will be conducted in 2 portions:

1. Enrollment A, which will consist of 2 treatment periods as follows and will be conducted in subjects with otomycosis:

   1. A randomized, double-blind, parallel-group treatment period. This treatment period will be referred to as the "Randomization Period" and will be followed by:
   2. An optional, open-label treatment period with miconazole oil. This treatment period will be referred to as the "Optional Open-label Extension."
2. Enrollment B will consist of open-label treatment with miconazole oil in subjects who will not be required to have signs and symptoms of otomycosis.

The study will start with Enrollment A, with an estimated 220 male or female subjects with otomycosis. Subjects will be randomly assigned in a 1:1 ratio to receive miconazole oil or vehicle (placebo), for 14 days. The study drug will be administered as 5 drops per ear at ~30 mg per drop instilled into the external ear canal of the ear(s) affected by otomycosis.

In the Randomization Period, both the subject and the investigator and study staff are blinded to the contents of the study drug.

At Screening/Baseline (Day 1), assessment of the signs and symptoms of otomycosis (pruritus, debris, visual examination for presence of fungal elements, and aural fullness), evaluation of medical history, pregnancy screening in female of childbearing potential, and, prior and concomitant medications, will be collected. Subjects with positive signs and symptoms of otomycosis and who meet all eligibility criteria will enter the study. Fungal culture of affected ear(s) will be taken, debris will be cleaned from the affected ear(s), and subject will be randomized and study drug dispensed. Treatment will be for 14 days. Day 8 On Treatment Visit will include clinical evaluation of otomycosis, cleaning of ear(s), and assessment of Adverse Events (AEs) and concomitant medications, and continue treatment up to Day 14. Day 15 End of Treatment Visit will include clinical evaluation of otomycosis and fungal culture, adverse events including Treatment emergent adverse events (TEAEs) and concomitant medications assessed. Day 22 Test of Cure Visit is an assessment of clinical signs and symptoms of otomycosis and fungal culture, AEs and concomitant medications assessed, and urine pregnancy test performed in women of childbearing potential.

Only the subjects that had positive fungal (mycological) culture at Baseline will be evaluated for efficacy. This is the Modified intent-to-treat (MITT) population.

The Optional Open-label Extension period will allow subjects to get miconazole oil for 14 days. No unblinding of the subject's treatment in the Randomization Period will occur at this time.

For Enrollment B, male or female subjects will be enrolled to receive miconazole oil to use for 14 days and will be evaluated for safety.

Intent-to-Treat (ITT) population are all subjects enrolled and randomized to treatment. Modified Intent-to-Treat (MITT) population are subjects in the ITT population with a clinical diagnosis of otomycosis confirmed by positive fungal culture at Baseline.

ELIGIBILITY:
Inclusion Criteria:

Randomized blinded initial phase of study:

* Male or non-pregnant, non-lactating females with a clinical diagnosis of uncomplicated otomycosis of the external ear only,
* Intact tympanic membrane in the ear(s) to be treated with study drug,
* In general good health as determined by medical examination and medical history,
* Free of clinically significant disease, including diabetes mellitus, that is not well-controlled or that could interfere with the study.

Open-label second phase of study:

* Male or non-pregnant, non-lactating females with an intact tympanic membrane in the ear(s) to be treated with study drug,
* In general good health as determined by medical examination and medical history,
* Free of clinically significant disease, including diabetes mellitus, that is not well-controlled or that could interfere with the study.

Exclusion Criteria::

* Presence of dermatoses or conditions of the ear that may interfere with evaluation of otomycosis or with safety evaluations, including concomitant otic infections that require antimicrobial treatment,
* Disease that has spread beyond the external ear(s), or pre-existing skin atrophy of the affected ear(s);
* Tympanostomy tube or perforated tympanic membrane;
* History of prior surgery directly affecting and compromising the external auditory canal and/or tympanic membrane, except for prior tympanostomy tube(s) that have already been removed and completely healed;
* Use of any topical medicated treatments for otomycosis within 14 days of study entry;
* Use of any systemic antifungal therapy within 28 days of study entry, warfarin within 28 days of study entry, immunosuppressive or immune-stimulating drugs within 28 days of study entry, or systemic steroids within 3 months of study entry;
* Fever of ≥100°F at study entry;
* Otomycosis that has been unresponsive to previous antifungal treatment;
* Known hypersensitivity to any of the components in the test formulation;
* Participation in another investigative trial within 28 days of study entry

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaldo Rivera, MD, Principal Investigator — University of Missouri-Columbia; Quyen T Nguyen, MD, Principal Investigator — UCSD; Kenneth Hodge, MD, Principal Investigator — Advanced ENT and Allergy; Patrick Dennis, MD, Principal Investigator — DelRicht Research; Sammy Vaught, MD, Principal Investigator — Lake ENT & FPS; Timothy Fitzgibbon, MD, Principal Investigator — OnSite Clinical Solutions; John Ansley, MD, Principal Investigator — Carolina ENT; Randall Ow, MD, Principal Investigator — DaVinci Research LLC; Oscar DeValle, MD, Principal Investigator — West Houston Clinical Research Service; Linda Woo, MD, Principal Investigator — Head and Neck Surgery Specialists; Brent Benscoter, MD, Principal Investigator — Sacramento ENT / DaVinci Research; Jeffrey Adelglass, MD, Principal Investigator — Research Your Health; Gary Brandt, MD, Principal Investigator — Delricht
Locations (12):
- United States (12):
  - Head and Neck Surgery Specialists, Chula Vista, California
  - UCSD, La Jolla, California
  - DaVinci Research, LLC, Roseville, California
  - Sacramento ENT / DaVinci Research, Sacramento, California
  - Lake ENT & FPS, Leesburg, Florida
  - Advanced ENT & Allergy, Louisville, Kentucky
  - DelRicht Research, New Orleans, Louisiana
  - University of Missouri, Columbia, Missouri
  - OnSite Clinical Solutions, Dillon, South Carolina
  - Carolina ENT, Orangeburg, South Carolina
  - West Houston Clinical Research Services, Houston, Texas
  - Research Your Health, Plano, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Treatment Arm: Participants randomized to Active Treatment with miconazole 2% oil, 5 drops into affected ear twice daily for 14 consecutive days
  miconazole 2% oil: Drug treatment of otomycosis for 14 days
- Placebo Treatment Arm: Participants randomized to Placebo Treatment (with vehicle oil placebo), 5 drops into affected ear twice daily for 14 consecutive days
  vehicle oil: Placebo treatment of otomycosis for 14 days
- Open-label Application Group: Application of miconazole 2% oil, 5 drops into each ear or the affected ear, twice daily for 14 consecutive days
  miconazole 2% oil: Drug application for 14 days
Period: Double-blind Treatment Period
Arm/Group | Active Treatment Arm | Placebo Treatment Arm | Open-label Application Group
Started | 89 | 90 | 0 (Open-label treatment group started under Period 2. Not applicable for Period 1.)
Completed | 84 | 79 | 0 (Open-label treatment group started under Period 2. Not applicable for Period 1.)
Not Completed | 5 | 11 | 0
Not completed — Adverse Event | 2 | 6 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — subject enrolled in the Optional Open Label arm | 0 | 1 | 0
Period: Enrollment B, Open Label Safety Group.
Arm/Group | Active Treatment Arm | Placebo Treatment Arm | Open-label Application Group
Started | 0 (Participants randomized to Active-treatment included in Period 1 only, double-blind randomized period.) | 0 (Participants randomized to Placebo-treatment included in Period 1 only, double-blind randomized period.) | 203 (Participants/subjects enrolled in open-label treatment arm were not required to have otomycosis, hence were not assessed for efficacy and not included in Period 1. This population was Not randomized, assessed only for safety, and included in Period 2 only.)
Completed | 0 | 0 | 203
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population - subjects enrolled and randomized according to treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment Arm | Placebo Treatment Arm | Open-label Treatment Arm | Total
Number analyzed (Participants) | 89 | 90 | 203 | 382
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 6 | 10 | 17
  Between 18 and 65 years | 56 | 61 | 178 | 295
  >=65 years | 32 | 23 | 15 | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 44 | 142 | 224
  Male | 51 | 46 | 61 | 158
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 19 | 38 | 80
  Not Hispanic or Latino | 66 | 71 | 165 | 302
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 2 | 6 | 6 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 12 | 49 | 68
  White | 76 | 68 | 133 | 277
  More than one race | 4 | 4 | 14 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Mycological culture [Count of Participants; unit: Participants]
  positive culture | 67 | 64 | 0 | 131
  negative culture | 22 | 26 | 0 | 48
  not cultured | 0 | 0 | 203 | 203
Otomycosis signs/symptoms - Pruritus [Count of Participants; unit: Participants]
  none | 1 | 2 | 0 | 3
  mild | 18 | 19 | 0 | 37
  moderate | 58 | 56 | 0 | 114
  severe | 12 | 13 | 0 | 25
  not assessed | 0 | 0 | 203 | 203
Otomycosis signs/symptoms - Debris [Count of Participants; unit: Participants]
  none | 0 | 0 | 0 | 0
  scant | 6 | 2 | 0 | 8
  moderate | 44 | 59 | 0 | 103
  heavy | 39 | 29 | 0 | 68
  not assessed | 0 | 0 | 203 | 203
Otomycosis signs/symptoms - Fungal elements [Count of Participants; unit: Participants]
  present | 89 | 90 | 0 | 179
  absent | 0 | 0 | 0 | 0
  not assessed | 0 | 0 | 203 | 203
Otomycosis signs/symptoms - Aural fullness [Count of Participants; unit: Participants]
  none | 0 | 1 | 0 | 1
  mild | 27 | 31 | 0 | 58
  moderate | 55 | 44 | 0 | 99
  severe | 7 | 14 | 0 | 21
  not assessed | 0 | 0 | 203 | 203

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Therapeutic Cure
Description: "therapeutic cure" is "mycological cure" plus "clinical cure, in the Modified intent to treat (MITT) only: patients with + fungal culture at baseline. Fungal culture results verified as (+) or (-) after enrollment.
  Intent to treat (ITT) population were all subjects enrolled and randomized. Active group: ITT=89 (100%), MITT=67 (75.3%); Placebo Group: ITT=90 (100%), MITT=64 (71.1%).
  Mycological cure is a negative mycological culture (culture is either positive or negative). Score=0 is best.
  Clinical cure is absence of all otomycosis signs and symptoms (s/s) of Pruritus, Debris, and Aural fullness, graded as (scores) 0=none, 1=mild, 2=moderate, 3=severe; and Presence of fungal elements, score 0=No fungal elements, 1=fungal elements present on visual inspection. Score=0 is best.
  Efficacy analysis was performed only on MITT (modified intent-to-treat) population, consisting of only those patients that had positive fungal culture at Baseline.
Time Frame: 21 days from first day of drug application
Population: MITT (modified intent-to-treat) population - only patients with positive mycological culture at Baseline. ITT (intent-to-treat) population were all subjects enrolled and randomized. Active group: ITT=89 (100%), MITT=67 (75.3%); Placebo Group: ITT=90 (100%), MITT=64 (71.1%).
Measure: Count of Participants; unit: Participants
Groups:
- Active Treatment Arm: Treatment with miconazole 2% oil, 5 drops into affected ear twice daily for 14 consecutive days
  miconazole 2% oil: Drug treatment of otomycosis for 14 days
- Placebo Treatment Arm: Treatment with the vehicle oil, placebo, 5 drops into affected ear twice daily for 14 consecutive days
  vehicle oil: Placebo treatment of otomycosis for 14 days
Arm/Group | Active Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 67 | 64
Participants
  Achieved Therapeutic cure (Score=0 fungal culture and clinical signs,symptoms) | 14 | 11
  Not Achieve Therapeutic cure (Positive fungal culture AND/OR clinical score 1 or greater each s/s | 53 | 53

2. Secondary Outcome: Percentage of Subjects With Mycological Cure
Description: Mycological cure is a negative mycological culture for the study ear at test of cure visit, in Modified intent to treat (MITT) only: patients with + fungal culture at baseline. Subjects that had negative fungal culture at Baseline were not included in MITT. Fungal culture results verified as (+) or (-) after enrollment.
  Grading is based on positive or negative mycological (fungal) culture. Negative culture is required.
  Efficacy analysis was performed only on MITT (modified intent-to-treat) population, consisting of only those patients that had positive fungal culture at Baseline.
  Intent to treat (ITT) population were all subjects enrolled and randomized. Active group: ITT=89 (100%), MITT=67 (75.3%); Placebo Group: ITT=90 (100%), MITT=64 (71.1%).
Time Frame: 21 days from first day of drug application
Population: MITT (modified intent-to-treat) population - only patients with positive mycological culture at Baseline. ITT population were all subjects enrolled and randomized. Active group: ITT=89 (100%), MITT=67 (75.3%); Placebo Group: ITT=90 (100%), MITT=64 (71.1%).
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 67 | 64
Participants
  Achieved mycological cure (negative fungal culture) | 24 | 15
  Not achieved mycological cure (positive fungal culture) | 43 | 49

3. Secondary Outcome: Percentage of Subjects With Clinical Cure
Description: Absence of all otomycosis signs and symptoms according to the scales for each individual sign/symptom. Score=0 is best.
  Clinical cure is absence of all otomycosis signs and symptoms of Pruritus, Debris, and Aural fullness, graded as (scores) 0=none, 1=mild, 2=moderate, 3=severe; and Presence of fungal elements, score 0=No fungal elements, 1=fungal elements present on visual inspection. Score=0 is best.
  Efficacy analysis was performed only on MITT (modified intent-to-treat) population, consisting of only those patients that had positive fungal culture at Baseline. Subjects that had negative fungal culture at Baseline were not included in MITT. Fungal culture results verified as (+) or (-) after enrollment.
  ITT (intent to treat) population were all subjects enrolled and randomized. Active group: ITT=89 (100%), MITT=67 (75.3%); Placebo Group: ITT=90 (100%), MITT=64 (71.1%).
Time Frame: 21 days from first day of drug application
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 67 | 64
Participants
  Achieved clinical cure (score = 0 for all signs, symptoms) | 22 | 14
  Not achieved clinical cure (score equal to or greater than 1 for each sign, symptom). | 45 | 50

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) are collected at the start and during use of study drug, Day 1 to Day 14 of study drug application. Collection of adverse events start the day the patient first applied the study drug and end the day of the patient's last study visit, Day 21. Adverse events were monitored through study completion.
Description: Treatment-emergent adverse events (TEAEs) are those with an onset on or after the date of first study drug application, up to the last application day for each patient. Adverse events were monitored through study completion.
Arm/Group | Active Treatment Arm | Placebo Treatment Arm | Open-label Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/90 | 0/203
Serious Adverse Events (participants affected / at risk) | 1/89 | 0/90 | 0/203
Other Adverse Events (participants affected / at risk) | 41/89 | 51/90 | 9/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment Arm (N=89) | Placebo Treatment Arm (N=90) | Open-label Treatment Arm (N=203)
acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — Acute kidney injury on Chronic Kidney Disease (CKD)
hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) — Hypotension
OTHER ADVERSE EVENTS (reported when occurring in more than 1.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment Arm (N=89) | Placebo Treatment Arm (N=90) | Open-label Treatment Arm (N=203)
ear discomfort (Ear and labyrinth disorders) | 8 (8) | 9 (9) | 0 (0)
vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 1 (1)
tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
ear infection fungal (Infections and infestations) | 27 (27) | 33 (33) | 0 (0)
otitis externa (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
otitis externa bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
otitis externa fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
application site irritation (General disorders) | 1 (1) | 0 (0) | 1 (1)
application site pain (General disorders) | 4 (4) | 3 (3) | 0 (0)
application site pruritus (General disorders) | 7 (7) | 8 (8) | 3 (3)
exposure to SARS-CoV-2 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
hypovolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The limited number of patients with otomycosis at any one time, and the lack of standardized FDA-approved clinical studies on otomycosis have proven to be challenging and difficult to assign predetermined analysis endpoints. This is in line with the challenges described in the FDA Accelerating Rare disease Cures Program, such as challenges faced when using well-established trial designs, and complexities in endpoint selection when there is limited information or understanding of the disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Proprietary Information will need prior written consent of the sponsor. PI will hold in confidence and not disclose any Proprietary Information unless disclosure has its prior written consent from sponsor, or that the information is disclosed to personnel who need to know. Sponsor will not prohibit PI to comply with applicable laws and regulations, provided PI gives prior written notice to Sponsor. Disclosure allowed if legally required and accorded confidential treatment.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT04432376/Prot_SAP_001.pdf